CLINICAL TRIAL: NCT05629858
Title: Time Restricted Eating for the Treatment of Polycystic Ovarian Syndrome (PCOS)
Brief Title: Time Restricted Eating for the Treatment of PCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Krista Varady, Professor of Nutrition, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-1500
Record Dates: First submitted 2022-11-17; First posted 2022-11-29 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Polycystic Ovary Syndrome; Obesity; Overweight
MeSH Terms: conditions — Polycystic Ovary Syndrome; Obesity; Overweight | interventions — Caloric Restriction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 6-hour Time restricted eating (TRE) (Experimental): Ad libitum food intake from 1-7 pm every day Fasting from 7-1 pm every day (18-h fast)
  Interventions: Other: 6-h Time restricted eating (TRE)
- Calorie restriction (CR) (Experimental): 25% energy restriction every day
  Interventions: Other: Calorie restriction (CR)
- Control (Experimental): Usual diet, eating over >10 h per day
  Interventions: Other: Control

INTERVENTIONS:
Other: 6-h Time restricted eating (TRE) — Ad libitum food intake from 1-7 pm every day Fasting from 7-1 pm every day (18-h fast)
  Arms: 6-hour Time restricted eating (TRE)
Other: Calorie restriction (CR) — 25% energy restriction every day
  Arms: Calorie restriction (CR)
Other: Control — Usual diet, eating over >10 h per day
  Arms: Control

SUMMARY:
BACKGROUND:

Polycystic ovary syndrome (PCOS) is the most common cause of anovulatory infertility among young women. This syndrome is a reproductive and endocrinological disorder that affects up to 18% of reproductive-aged women. To date, the only strategy shown to reverse PCOS is sustained weight loss of 5-10%. At present, daily calorie restriction (CR) is the main diet prescribed to patients with PCOS for weight loss. However, some women find it difficult to adhere to CR because calorie intake must be vigilantly monitored every day. Considering these problems with CR, another approach that limits timing of food intake, instead of number of calories consumed, has been developed. This diet is called "time restricted eating" (TRE) and involves confining the period of food intake to 6-8 h per day. TRE allows individuals to self-select foods and eat ad libitum during a large part of the day, which can increase compliance to these protocols. Recent findings show that TRE significantly reduces body weight and insulin resistance in adults with obesity. However, no randomized controlled trials have studied the role of TRE in treating PCOS.

OBJECTIVE:

We conducted a 6-month, randomized, controlled trial comparing the effects of 6-h TRE (eating all food between 1:00 pm to 7:00 pm, without calorie counting), versus CR (25% energy restriction daily), and a control group (eating over a period of 10 or more hours per day), on body weight and PCOS symptoms in a racially-ethnically diverse group of females with PCOS.

METHODS:

A 6-month randomized, controlled, parallel-arm trial will be implemented. Females with overweight/obesity and PCOS will be randomized to 1 of 3 groups: (1) 6-h TRE (eating all food between 1:00 pm to 7:00 pm, without calorie counting); (2) CR (25% energy restriction daily); or (3) control group (eating over a period of 10 or more hours per day).

ELIGIBILITY:
4.1 Inclusion criteria:

* Diagnosed with PCOS based on the Rotterdam criteria in which two of three of the following criteria are present: (i) androgen excess skin manifestations (hirsutism, acne, and seborrhea) and/or hyperandrogenemia (total testosterone >55 pg/ml, free testosterone >9.4 pg/ml, androstenedione >2.1 ng/ml or DHEA-S >340 ug/dl); (ii) polycystic ovarian morphology on ultrasound (ovarian volume >10 cc and /or antral follicle count 20 in at least one ovary); and (iii) chronic oligo-amenorrhea (intermenstrual intervals >35 days or 7 periods/year)
* BMI between 25-50 kg/m2
* Age between 18-45 years

4.2 Exclusion criteria:

* Postmenopausal (absence of menses for >2 y)
* Diagnosed type 1 diabetes or type 2 diabetes
* Previously diagnosed with a mood depressive disorder (by a doctor or psychologist)
* Have a history of eating disorders (anorexia, bulimia, or binge eating disorder)
* Are not weight stable for 3 months prior to the beginning of the study
* Are taking drugs that affect study outcomes, such as oral contraceptives, weight loss, insulin-sensitizing agents, androgen antagonists, anti-seizure, or antipsychotic medication (within 2 months of starting study)
* Are currently following a TRE protocol
* Are athletes or those engaging in >1 hour of high-intensity training on more than 5 days/week
* Are active smokers (within 3 months of starting the study)
* Do not have a Wi-Fi connection at home (needed for zoom calls)
* Pregnant or trying to become pregnant

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women with PCOS and overweight or obesity will be invited to participate in the study.
Enrollment: 76 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Change in percent body weight | Measured at month 0 and 6
  Measured by an electronic scale

SECONDARY OUTCOMES:
Change in fat mass, lean mass, visceral fat mass | Measured at month 0 and 6
  Measured by DXA
Change in waist circumference | Measured at month 0 and 6
  Measured by a measuring tape
Change in insulin resistance | Measured at month 0 and 6
  Measured by HOMA-IR (Homeostatic Model Assessment for Insulin Resistance)
Change in insulin sensitivity | Measured at month 0 and 6
  Measured by QUICKI (Quantitative insulin sensitivity check index)
Change in fasting glucose | Measured at month 0 and 6
  Measured by a commercial lab (Medstar, IL)
Change in fasting insulin | Measured at month 0 and 6
  Measured by a commercial lab (Medstar, IL)
Change in HbA1c | Measured at month 0 and 6
  Measured by a commercial lab (Medstar, IL)
Change in blood pressure | Measured at month 0 and 6
  Measured by a blood pressure cuff
Change in heart rate | Measured at month 0 and 6
  Measured by a blood pressure cuff
Change in plasma lipids (LDL cholesterol, HDL cholesterol, triglycerides) | Measured at month 0 and 6
  Measured by a commercial lab (Medstar, IL)
Change in reproductive hormones (testosterone, DHEA, SHBG) | Measured at month 0 and 6
  Measured by a commercial lab (Medstar, IL)
Change in free androgen index (FAI) | Measured at month 0 and 6
  FAI is calculated by multiplying total testosterone by 100 and dividing by sex hormone binding globulin (SHBG)
Change in energy and nutrient intake | Measured at month 0 and 6
  Measured by 7-day food record
Change in dietary adherence | Measured at month 0 and 6
  Measured by survey
Change in physical activity (steps/d) | Measured at month 0 and 6
  Measured by pedometer
Change in PCOS symptoms | Measured at month 0 and 6
  Measured by a validated questionnaire (PMSIS: Premenstrual symptom impact survey)
Change in hirsutism | Measured at month 0 and 6
  Measured by a validated questionnaire (mFG: modified Ferriman-Gallwey hirsutism scale)
Change in acne severity | Measured at month 0 and 6
  Measured by a validated questionnaire (CASS: Comprehensive acne severity scale)
Change in seborrhea | Measured at month 0 and 6
  Measured by clinical assessment
Change in menstrual regularity and blood loss | Measured at month 0 and 6
  Measured by survey (PBAC: Pictorial blood loss assessment chart)
Occurences of adverse events | Measured at month 0 and 6
  Measured by adverse event survey

CONTACTS AND LOCATIONS:
Overall Officials: Krista Varady, PhD, Principal Investigator — University of Illinois Chicago
Locations (1):
- University of Illinois Chicago, Chicago, Illinois, United States